CLINICAL TRIAL: NCT07077850
Title: The Effectiveness of Intravenous Dexamethasone Prophylaxis in Preventing Post-operative Urinary Retention in Spinal Anesthesia at Al-Makassed Hospital
Brief Title: Effect of IV Dexamethasone on Post-op Urinary Retention After Spinal Anesthesia
Acronym: DEX-PUR
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Quds University (Other)
Responsible Party: Principal Investigator, Abeer Hasan, Abeer Jafar Dar Hasan , General Surgery Senior Resident, MBBS, Al-Quds University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: DEX-PUR Trial
Record Dates: First submitted 2025-07-12; First posted 2025-07-22 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Post Operative Urinary Retention; Spinal Aneshtesia
Keywords: POUR; Spinal Anesthesia; Dexamethasone; Intravenous Corticosteriods; Urinary Complications; Perioperative Complications; Placebo-Controlled Trial; Randomized Controlled Trial; Al-Makassed Hospital; Postoperative Urinary Retention
MeSH Terms: interventions — Dexamethasone; dexamethasone 21-phosphate; Saline Solution; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned in a 1:1 ratio to receive either a single 8 mg dose of intravenous dexamethasone or a placebo (0.9% normal saline) prior to surgery under spinal anesthesia. Each participant remains in their assigned group throughout the study.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This is a double-blinded study. Both participants and outcome assessors are unaware of the group assignments. A non-participating physician performed the randomization using a computer-generated block randomization list. Study drugs (dexamethasone or placebo) are prepared in identical syringes labeled with participant codes only, ensuring that care providers and investigators remain blinded during the intervention and follow-up period.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm 2: Placebo Group (Participants receiving intravenous 0.9% saline as placebo) (Placebo Comparator): Participants in this arm will receive an intravenous injection of 0.9% normal saline (placebo) before undergoing surgery under spinal anesthesia. This group is used to compare the effect of dexamethasone on the incidence of postoperative urinary retention (POUR).
  Interventions: Drug: Normal Saline (0.9% NaCl)
- Arm 1: Dexamethasone group (Experimental): Participants in this arm will receive a single 8 mg dose of intravenous dexamethasone before undergoing surgery under spinal anesthesia. The intervention is administered preoperatively to evaluate its effectiveness in reducing the risk of postoperative urinary retention (POUR).
  Interventions: Drug: Dexamethasone (IV)

INTERVENTIONS:
Drug: Dexamethasone (IV) — Intravenous administration of 8 mg dexamethasone sodium phosphate given as a single dose before surgery under spinal anesthesia. This corticosteroid is being evaluated for its potential to prevent postoperative urinary retention (POUR) by reducing inflammation and other perioperative effects.
  Other Names: Dexamethasone Sodium Phosphate
  Arms: Arm 1: Dexamethasone group
Drug: Normal Saline (0.9% NaCl) — Intravenous administration of 0.9% normal saline (placebo) given as a single dose before surgery under spinal anesthesia. This inert solution is used to compare against the active drug dexamethasone to determine its effect on postoperative urinary retention (POUR).
  Other Names: Isotonic Saline
  Arms: Arm 2: Placebo Group (Participants receiving intravenous 0.9% saline as placebo)

SUMMARY:
What is this study about? This study is testing whether a common medication called dexamethasone, given through a vein (IV) before surgery, can help prevent a problem called postoperative urinary retention (POUR). POUR means having trouble urinating after surgery, which can cause discomfort and sometimes requires using a catheter.

Who can join the study? The study includes adult People who are having surgery with spinal anesthesia at Al-Makassed Hospital. People who have certain medical conditions, use steroids regularly, or need a catheter during surgery cannot join.

What will happen in the study?

Participants will be randomly assigned to one of two groups:

* One group will get 8 mg of IV dexamethasone before surgery.
* The other group will get a saltwater (placebo) injection. Neither the participants nor the doctors will know which treatment they receive.

After surgery, the researchers will check how soon each participant can urinate and whether they need a catheter.

Why is this study important? POUR can slow recovery and cause complications. Dexamethasone is already used for other reasons like nausea and swelling. This study will help find out if it also lowers the risk of POUR in people getting spinal anesthesia.

DETAILED DESCRIPTION:
Postoperative urinary retention (POUR) is a common complication following spinal anesthesia, affecting patient comfort, recovery, and sometimes requiring catheterization. While dexamethasone is routinely used to prevent nausea and inflammation in surgical patients, its potential role in preventing POUR has not been fully explored, especially in the context of spinal anesthesia.

This study is a prospective, randomized, double-blind, placebo-controlled clinical trial conducted at Al-Makassed Hospital. It aims to evaluate whether a single preoperative intravenous dose of 8 mg dexamethasone reduces the incidence of POUR in adult patients undergoing elective surgery under spinal anesthesia.

Eligible participants are randomized into two equal groups using block randomization. One group receives 8 mg of IV dexamethasone, and the other receives a placebo (0.9% saline). Both patients and assessors are blinded to group assignment. Data will be collected on age, BMI, comorbidities (including history of BPH or prior POUR), current anticholinergic drug use, anesthetic agent and dose, which level of spinal anesthesia (e.g. L3-L4), type of surgery, IV fluid volume, and duration of operation.

The primary outcome is the incidence of POUR, defined as failure to void within 6 hours after surgery and requiring catheterization. Secondary outcomes include time to first void and the overall need for urinary catheterization. Safety data will also be recorded, and any adverse events related to dexamethasone will be reported.

The study has been approved by the Al-Quds University Research Ethics Committee. All participants will provide informed consent prior to enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients at Al-Makassed Hospital undergoing spinal anesthesia for surgery

Exclusion Criteria:

* Chronic steroid use
* Individuals who should not be administered dexamethasone
* Have a history of urological issues or procedures
* Have neurological disorders
* Using an intraoperative Foley's catheter
* Operations for possible nerve damage

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1084 (Actual)
Dates: Start 2025-08-20 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-08-20 (Estimated)

PRIMARY OUTCOMES:
Incidence of Postoperative Urinary Retention (POUR) | Measured within 6 hours postoperatively.
  The percentage of participants who fail to void within 6 hours after surgery and require urinary catheterization.

SECONDARY OUTCOMES:
Time to First Urination | Recorded within the first 24 hours after surgery.
  Time elapsed from the end of surgery until the participant first voids spontaneously.
Need for Urinary Catheterization | During hospital stay post-surgery (up to 24 hours)
  Number and percentage of participants who require catheterization at any time during postoperative monitoring.
Adverse Events Related to Dexamethasone | From drug administration to 24 hours postoperative.
  Incidence and type of adverse events possibly related to dexamethasone administration (e.g., allergic reactions).

CONTACTS AND LOCATIONS:
Overall Officials: Abeer J Dar Hasan, MD, Principal Investigator — Al-Makassed Islamic Charitable Society Hospital and Al-Quds University; Mohammed M Maree, MD, Study Director — Al-Makassed Islamic Charitable Society Hospital and Al-Quds University
Locations (1):
- Al-Makassed Islamic Charitable Society Hospital, East Jerusalem, Al-Makassed Islamic Charitable Society Hospital, Palestinian Territories

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared because this study is conducted at a single center with limited infrastructure for data sharing. Additionally, the current ethical approval and informed consent do not include provisions for sharing de-identified participant-level data with external researchers.

REFERENCES:
- [Background] Neff SP, Stapelberg F, Warmington A. Excruciating perineal pain after intravenous dexamethasone. Anaesth Intensive Care. 2002 Jun;30(3):370-1. doi: 10.1177/0310057X0203000319. PMID 12075649
- [Background] Toftegaard M, Knudsen F. Massive vasopressin-resistant polyuria induced by dexamethasone. Intensive Care Med. 1995 Mar;21(3):238-40. doi: 10.1007/BF01701480. PMID 7790612
- [Background] Primack A, Kajubi S. Insulin and growth hormone response to an oral glucose load in Ugandan hepatocellular carcinoma patients. East Afr Med J. 1974 Aug;51(8):574-8. No abstract available. PMID 4371198
- [Background] Denham M, Donovan K, Wetoska N, Kuchta K, Carbray J, Linn JG, Denham W, Haggerty SP, Joehl R, Ujiki M. Effects of dexamethasone on postoperative urinary retention after laparoscopic inguinal hernia repair. Surg Endosc. 2019 Sep;33(9):3008-3013. doi: 10.1007/s00464-018-6572-7. Epub 2018 Nov 7. PMID 30406386
- [Background] Splinter WM, Roberts DJ. Dexamethasone decreases vomiting by children after tonsillectomy. Anesth Analg. 1996 Nov;83(5):913-6. doi: 10.1097/00000539-199611000-00004. PMID 8895262
- [Background] Levin RM, Longhurst PA, Monson FC, Kato K, Wein AJ. Effect of bladder outlet obstruction on the morphology, physiology, and pharmacology of the bladder. Prostate Suppl. 1990;3:9-26. doi: 10.1002/pros.2990170503. PMID 1689174
- [Background] Kamphuis ET, Ionescu TI, Kuipers PW, de Gier J, van Venrooij GE, Boon TA. Recovery of storage and emptying functions of the urinary bladder after spinal anesthesia with lidocaine and with bupivacaine in men. Anesthesiology. 1998 Feb;88(2):310-6. doi: 10.1097/00000542-199802000-00007. PMID 9477049

DOCUMENTS (4):
  • Study Protocol and Statistical Analysis Plan: Proposal (2025-07-01): https://cdn.clinicaltrials.gov/large-docs/50/NCT07077850/Prot_SAP_000.pdf
  • Study Protocol and Statistical Analysis Plan: application form (2025-07-01): https://cdn.clinicaltrials.gov/large-docs/50/NCT07077850/Prot_SAP_001.pdf
  • Study Protocol and Statistical Analysis Plan: check list (2025-07-01): https://cdn.clinicaltrials.gov/large-docs/50/NCT07077850/Prot_SAP_002.pdf
  • Study Protocol and Statistical Analysis Plan: REC approval (2025-07-01): https://cdn.clinicaltrials.gov/large-docs/50/NCT07077850/Prot_SAP_003.pdf